CLINICAL TRIAL: NCT05798832
Title: Evaluation of Virtual Reality and Traditional Training in Basic Life Support Training: The Case of Paramedic Student Group
Brief Title: An Evaluation of Virtual Reality and Traditional Training in Basic Life Support Training
Acronym: VR-BLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Derya Aslan Huyar, Lecturer, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BursaU
Record Dates: First submitted 2023-02-19; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Education; Virtual Reality; Basic Cardiac Life Support
Keywords: Virtual Reality, Educational; Basic Cardiac Life Support

STUDY DESIGN:
Intervention Model Description: An experimental and a pretest-posttest control group design method were applied in this regard.
Who Masked: Outcomes Assessor
Masking Description: The person who will make the statistical analysis; He does not know which group the participants in our study belong to and he does not know the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): The active control group was given traditional Basic Life Support, which already practiced in most schools.For the traditional BLS training group; basic life support was given a lesson in the classroom for 45 to 50 minutes, demonstrated on a model, and the training session was ended after a question and answer session. In terms of standardization of the trainings, the trainings were given by Derya ASLAN HUYAR.
  Interventions: Other: Traditional training group
- experimental (Experimental): Basic Life Support training with VR was given to the experimental group.For the VR BLS training group; The use of VR was introduced in the VR hall. The lexical meanings of the basic concepts of BLS were explained. The student received training on a scenario he chose in the training module, and then he was asked to perform the steps individually in the assessment mode. After the training was completed, a question-answer was made and the session was closed. In terms of standardization of the trainings, the trainings were made by Derya ASLAN HUYAR.
  Interventions: Other: Virtually reality training group

INTERVENTIONS:
Other: Virtually reality training group — BLS Training with VR
  Arms: experimental
Other: Traditional training group — BLS Training with Traditional
  Arms: Active Comparator

SUMMARY:
type of study:A parallel-group trial design was used.

The main question[s] it aims to answer are:

1. HI; The "Basic Life Support Knowledge Assessment Form" score average of the students in the intervention group participating in the VR will be higher than the control group.
2. H1; The Basic Life Support Application Evaluation Form score average of the students in the intervention group participating in the VR will be higher than the control group.

A. For the classical BLS training group; Traditional BLS VR Training will be held in the classroom environment for 45 minutes in the form of a lecture, the training session will be terminated after watching the video and answering questions. Trainings will be conducted by Derya ASLAN HUYAR in terms of standardization of trainings.

B.For VR BLS training group; After the introduction of VR in the VR hall, after the explanation of the basic concepts of BLS and the completion of the training through VR BLS scenarios, question-answer will be made and the session will be closed. Trainings will be conducted by Derya ASLAN HUYAR in terms of standardization of trainings.

DETAILED DESCRIPTION:
An experimental and a pretest-posttest control group design method were applied in this regard.

Population and Sample: The population of the research consists of 89 paramedic students studying in the first grade of the Bursa Uludag University First and Emergency Aid Program in the spring semester of the 2021-2022 academic year.The sample size was determined by means of a power analysis.When the effect size of the difference in knowledge levels between the two groups at 80% power and 5% significance level is taken as 0.70, 34 participants in each group are required, with a total of 68 participants.They were randomly assigned to the experimental and control groups.Participants; Being a first-year paramedic student, not having received basic life support training, and voluntarily agreeing to participate in the study were determined as inclusion criteria.

The number of people to be sampled from the universe was determined by power analysis. When the effect size of the difference in knowledge levels between the two groups at 80% power and 5% significance level is taken as 0.70, 34 participants in each group are required, with a total of 68 participants.

Participants will be assigned to the experimental and control groups by randomization. Participants; Being a first-year paramedic student, not having received basic life support training, and voluntarily agreeing to participate in the study were determined as inclusion criteria.

Data Collection Tools Created by researchers; The "Descriptive Information Form" consists of 6 items. (Annex 6-5) "Basic Life Support Information Evaluation Form" was developed by Tank. This form, which consists of 10 multiple-choice questions, adapted according to the Critical Skills Descriptors of the Adult Cardiopulmonary Resuscitation and Automatic External Defibrillator Skills Test published by the American Heart Association; questions their level of knowledge about basic life support application. Each correct answer given by the student in the form will be evaluated as 1 point and the average score will be calculated. Students will be able to get a minimum of 0 and a maximum of 10 points (Appendix 6-5) "Basic Life Support Application Evaluation Form" was developed by Tank , it consists of 20 items. This form is used to evaluate the participant's skill status during BLS practice. In the form containing the application steps, the student's ability to perform the application will be evaluated as 1 point for each correct step, and the average score will be calculated. The participant will be able to get a minimum of 0 and a maximum of 20 points at the end of the evaluation of the 20-item form. (Annex 6-5) Data Analysis: SPSS package program will be used.

Research Flow Process:

Basic Life Support (BLS) Virtual Reality (VR) and Basic Life Support Traditional Education Program Flow Process Steps

1. Pre-Training Evaluation Students randomly assigned to the VR and Classical education group; "Descriptive Information Form" and "Basic Life Support Information Evaluation Form" will be filled.
2. Education

   1. For the classical BLS training group; Traditional BLS VR Training will be held in the classroom environment in the form of lectures for 45 minutes, and the training session will end after watching the video and question and answering. In terms of standardization of the trainings, the trainings will be given by Derya ASLAN HUYAR.
   2. For the VR BLS training group; After the VR presentation in the VR hall, after the explanation of the basic concepts of BLS and the completion of the training on VR BLS scenarios, there will be a question and answer session and the session will be closed. In terms of standardization of the trainings, the trainings will be given by Derya ASLAN HUYAR.
3. Initial Evaluation After Training For practices, students will be divided into groups of 6 to 8 people.

   1. Med-Sim Training simulator will be introduced by the Training Coach and BLS application steps will be demonstrated.
   2. A BLS scenario will be given to the participants in the classical and VR BLS training groups. Then, each participant will perform the application steps on the Med-Sim simulation model. In the meantime, each participant will be evaluated in terms of skills by using the "Basic Life Support Application Evaluation Form" by Derya ASLAN HUYAR and Yeliz ŞAPULU ALAKAN.
   3. Participants in the Classical and VR BLS training groups will fill out the "Basic Life Support Information Evaluation Form" after the training.
4. Second Evaluation After Training One month after the training, just like in the phases applied in the first measurement; BLS scenario will be given to the participants in both classical and BLS training groups. Each participant will be evaluated in terms of skills by Derya ASLAN HUYAR and Yeliz ŞAPULU ALAKAN using the "Basic Life Support Application Evaluation Form" while the participants are doing the application steps on the Med-Sim simulation model.

   One month after the training, the participants in the Classic and VR BLS training groups will fill out the "Basic Life Support Information Evaluation Form" after the training.
5. Third Evaluation After Training Planned steps in other measurements will be followed in the same way. Three months after the training, the participants in the Classical and BLS training groups will be given a BLS scenario and asked to do the application steps on the Med-Sim simulation model. Meanwhile, each participant will be evaluated in terms of skills by using the "Basic Life Support Application Evaluation Form" by Derya ASLAN HUYAR and Yeliz ŞAPULU ALAKAN while the participants are doing the application steps on the Med-Sim simulation model.

Three months after the training, the participants in the Classic and VR BLS training groups will fill out the "Basic Life Support Information Evaluation Form" after the training.

ELIGIBILITY:
Inclusion Criteria:

* Being a first-year paramedic student,
* not having received basic life support training
* voluntarily agreeing to participate in the research,

Exclusion Criteria:

* have previous BLS training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
before the intervention | via google form. Before the intervention
  Before the training of the experimental and control group participants, BLS knowledge was measured."Basic Life Support Information Evaluation Form" is organized according to the Adult Cardiopulmonary Resuscitation and Automatic External Defibrillator Skill steps published by the American Heart Association and consists of 10 multiple choice questions.
  Each correct answer is 1 point. minimum 0, maximum 10 points can be scored.

SECONDARY OUTCOMES:
immediately after the intervention, | via google form. it took a total of 2 weeks to complete the skill measurements of the control and experimental groups. Control group: May 16-20 experimental group may 23-27
  The BLS knowledge level of the experimental and control groups was measured with the questionnaire.
  In addition, the researchers gave each student an appointment individually so that the skill levels of both groups could be measured. "Basic Life Support Application Evaluation Form" consists of 20 items. In the form containing the application steps, 1 point is taken for each correct step. The participant will be able to get a minimum of 0 and a maximum of 20 points.
  The researchers asked the participants to apply the BLS steps on the BLS model. The researchers marked their observations as checklist. Each student was given feedback after the application.
1st months after the intervention. | via google form. It took a total of 2 weeks to complete the skill measurements of the control and experimental groups. Control group: 20-24 June experimental group: 27 June 1 July
  The BLS knowledge level of the experimental and control groups was measured with the questionnaire.
  In addition, the researchers gave each student an appointment individually so that the skill levels of both groups could be measured. "Basic Life Support Application Evaluation Form" consists of 20 items. In the form containing the application steps, 1 point is taken for each correct step. The participant will be able to get a minimum of 0 and a maximum of 20 points.
  The researchers asked the participants to apply the BLS steps on the BLS model. The researchers marked their observations as checklist. Each student was given feedback after the application.
3rd months after the intervention. | via google form. Each student was given an appointment to assess the students' BLS skill level. It took a total of 2 weeks to complete the skill measurements of the control and experimental groups.19 -23 Sep.]
  The BLS knowledge level of the experimental and control groups was measured with the questionnaire.
  In addition, the researchers gave each student an appointment individually so that the skill levels of both groups could be measured. "Basic Life Support Application Evaluation Form" consists of 20 items. In the form containing the application steps, 1 point is taken for each correct step. The participant will be able to get a minimum of 0 and a maximum of 20 points.
  The researchers asked the participants to apply the BLS steps on the BLS model. The researchers marked their observations as checklist. Each student was given feedback after the application.

CONTACTS AND LOCATIONS:
Overall Officials: derya aslan huyar, Principal Investigator — Bursa Uludag Universty
Locations (1):
- Bursa Uludağ Üniversitesi, Bursa, Nilüfer, Turkey (Türkiye)